CLINICAL TRIAL: NCT00069550
Title: Pathogenesis of Rett Syndrome: Natural History and Treatment
Brief Title: Independent Studies of Dextromethorphan and of Donepezil Hydrochloride for Rett Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HD024448; 5P01HD024448 (NIH)
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-12

CONDITIONS: Rett Syndrome
Keywords: Glutamate/NMDA receptors; Cholinergic upregulation; Dextromethorphan; Donepezil hydrochloride; Aricept
MeSH Terms: conditions — Rett Syndrome | interventions — Dextromethorphan; Donepezil

INTERVENTIONS:
Drug: dextromethorphan
Drug: donepezil hydrochloride

SUMMARY:
Rett syndrome (RTT) is a disorder in which the nervous system does not develop properly. RTT generally affects girls, but there are some boys who have been diagnosed with RTT. Symptoms of RTT include small brain size, poor language skills, repetitive hand movements, and seizures. This study will evaluate the effectiveness of two drugs in treating the symptoms of RTT.

DETAILED DESCRIPTION:
RTT is a neurodevelopmental disorder characterized by apparently normal early development followed by loss of purposeful hand use, distinctive hand stereotypies, slowed brain growth, loss of language, respiratory irregularities, GI disturbances, gait abnormalities, seizures, and mental retardation. These symptoms appear between ages 6 and 18 months (stage 2 of the disease) following apparently normal development (stage 1). Subsequently, there is gradual stabilization of severe mental retardation and motor compromise (stage 3). The majority (70% to 80%) of patients demonstrate mutations in the methyl-CpG-binding-protein-2 (MeCP2) gene, a transcription repressor located on chromosome Xq28. The disorder predominantly affects females, but a few males with mutations in MeCP2 have been identified, even though many of them do not have the classic symptoms recognized in females.

Recent studies demonstrate increased brain N-methyl-D-aspartate (NMDA) receptors in stages 2 and 3 of the disease. This age-specific increase in glutamate levels and their receptors contribute to brain damage. This first study will examine the effectiveness of dextromethorphan, an NMDA receptor antagonist, to ameliorate symptoms. Participants will be randomized to receive one of three doses of dextromethorphan. All participants will be admitted to the hospital for three days at the beginning of the study. During the hospitalization, participants will undergo physical exam, Dexascan, MRI, EEG, behavioral assessment, laboratory testing, and neuropsychological evaluations. Six months after baseline assessment, participants will be rehospitalized for 3 days for similar assessments.

Reduction in choline acetyltransferase activity in RTT patients may also contribute to disturbed cortical development and psychomotor retardation in RTT. Therefore, the second part of the study will evaluate the effect of donepezil hydrochloride, an inhibitor of acetylcholine-esterase, on acetylcholine levels. This portion of the study will not begin until pharmacokinetic data for donepezil in children is available.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Rett syndrome
* Mutation in MeCP2 gene
* Typical EEG abnormalities (disorganized background, frontal central spikes, rhythmic theta)

Exclusion Criteria

* Features of Rett syndrome with absence of MeCP2 mutation
* Non-specific EEG changes

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2004-09; Study Completion 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: SakkuBai R. Naidu, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States